CLINICAL TRIAL: NCT01695096
Title: High Versus Free Humidity Incubators; A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Ganna Hospital (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Laboratory Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ibnsinaH; ibnsinaH (Other: ibnsinaH)
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Ongoing Pregnancy Rate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The Embryos will be cultured on a humidity free incubator (Experimental): We will set the humidity level to 0.0% in the IVF incubator that will be used for culturing the Human embryos after ICSI procedure and we will monitor the outcome embryologically and clinically and record the results.
  Interventions: Other: The Embryos will be cultured on a humidity free incubator
- The Embryos will be cultured on a >95% humidity incubator (Placebo Comparator): We will set the humidity level to > 95% in the IVF incubator that will be used for culturing the Human embryos after ICSI procedure and we will monitor the outcome embryologically and clinically and record the results.
  Interventions: Other: The Embryos will be cultured on a >95% humidity incubator

INTERVENTIONS:
Other: The Embryos will be cultured on a humidity free incubator — We will set the humidity level to 0.0% in the IVF incubator that will be used for culturing the Human embryos after ICSI procedure and we will monitor the outcome embryologically and clinically and record the results.
  Arms: The Embryos will be cultured on a humidity free incubator
Other: The Embryos will be cultured on a >95% humidity incubator — We will set the humidity level to 95% in the IVF incubator that will be used for culturing the Human embryos after ICSI procedure and we will monitor the outcome embryologically and clinically and record the results.
  Arms: The Embryos will be cultured on a >95% humidity incubator

SUMMARY:
To compare Top quality embryos either day3 or day 5, Pregnancy rate and most importantly ongoing pregnancy rate between high humidity incubators and humidity free incubators

DETAILED DESCRIPTION:
When the IVF started the majority of incubators designed to support high humidity because the designers and IVF specialists believed that the humidity will maintain stable ph and Temp.

Recent reports suggest that humidity is recommended and the others suggest no difference So we decide to go for this RCT. Nevertheless; high humidity is maintained in vivo (uterus and fallopian tubes) due to the fluid content and stable body temperatures at 37°C. David McCulloch reported 15% reduction of the miscarriage rate after changing the humidity from 76% to 100% (Textbook of Assisted Reproductive Techniques: Laboratory Perspectives, Fourth Edition). Some embryologists claim that the humidity free incubators may increase the chance of chemical pregnancy and early fetal loss (Private center IbnSina IVF, Sohag, Egypt. unpublished data). This observations are never tested in a well designed randomized clinical trial (RCT) to eliminate the probability of chance and to reach a solid evidence.

The question that should be asked : is high humidity culture should be applied or there is no difference between dry and high humidity culture conditions?

ELIGIBILITY:
Inclusion Criteria:

* < 33 years, BMI<30,
* Normo Responder(>8 MII)
* Fresh Cycle
* Ist attempt
* Normal or mild oligoasthenoteratozoospermia.

Exclusion Criteria:

* Testicular sperm
* < 8 MII collected
* difficult transfer cycle
* Endometriotic patients
* Poor Endometrium < 8mm diameter at Ovum Pickup
* any other medical diseases

Ages: 18 Years to 33 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 284 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 18 months
  assessing the ongoing pregnancy rate and its difference between the 2 study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad F. Abdel-Raheem, Lab Director, Principal Investigator — IBNSINA IVF Center; Muhammad El Hady, Lab Director, Principal Investigator — Ganna Hospital; Mohamed Y. Abdel-Rahman, M.D., Study Director — IBNSINA IVF center
Locations (2):
- Egypt (2):
  - Gannah IVF unit, Gannah Hospital, Giza, Giza Governorate
  - IbnSina IVF unit, IbnSina Hospital, El Areef Square, Sohag, Sohag Governorate

REFERENCES:
- [Derived] Fawzy M, AbdelRahman MY, Zidan MH, Abdel Hafez FF, Abdelghafar H, Al-Inany H, Bedaiwy MA. Humid versus dry incubator: a prospective, randomized, controlled trial. Fertil Steril. 2017 Aug;108(2):277-283. doi: 10.1016/j.fertnstert.2017.05.036. Epub 2017 Jun 23. PMID 28651960
- See also: Facebook group for Gannah hospital, site doing the study — http://www.facebook.com/groups/314911565200565/